CLINICAL TRIAL: NCT06196476
Title: The Effectiveness of an Interactive Digital-based Educational Program in Unleashing Awareness, Self-Efficacy, and Environmental Activism in the Face of Climate Change Among Primary Health Care Rural Nurses: A Randomized Control Trial
Brief Title: Interactive Digital-based Educational Program and Climate Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hashem El-Monshed, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Climate Change MansU-Nursing
Record Dates: First submitted 2023-12-23; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Climate Change; Interactive Digital-based Educational Program; Rural Nurses
Keywords: Climate Change

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The participants in this group received routine nursing information in which the nurse discussed general knowledge of climate change awareness regarding the management of reducing Climate Anxiety effects to primary health care nurses.
- Intervention Group (Experimental): The participants in this group received an empowerment-based intervention in terms of interactive digital-based educational program regarding the promoting literacy, pro-environmental attitudes, self-efficacy, and reducing climate anxiety.
  The Interactive digital-based educational program Sessions:
  Session 1: The road start to green planet: Introductory to climate change concept Session 2: Towards Climate Change Literacy Modifications: remove the cover on illiteracy.
  Session 3: Green scrubs and green environment: raising climate activities and environment self-efficacy Session 4: Strengthen resilience to overcome climate related anxiety Session 5: Sustaining phase: closing session
  Interventions: Behavioral: Interactive digital-based educational program

INTERVENTIONS:
Behavioral: Interactive digital-based educational program — The Interactive digital-based educational program Sessions:
  Session 1: The road start to green planet: Introductory to climate change concept Session 2: Towards Climate Change Literacy Modifications: remove the cover on illiteracy.
  Session 3: Green scrubs and green environment: raising climate activities and environment self-efficacy Session 4: Strengthen resilience to overcome climate related anxiety Session 5: Sustaining phase: closing session
  Arms: Intervention Group

SUMMARY:
Nursing's climate action position may shift from a white and wealthy world to a more inclusive one. Nurses in Egypt and elsewhere have found resonance with this method of campaigning, pressing their employers to implement ambitious environmental regulations (Jones-Berry, 2019). Nursing should be open to utilizing its voice to effect change. Even when nurses recognize their obligation to assist in solving climatic and environmental challenges, many view it as secondary to other parts of their profession (Anker et al., 2015). Nurses who are concerned about sustainability must have the confidence to speak out, since actions such as modelling sustainable practices, pushing for change, advocating for community health, or criticizing prominent organizations may make nurses unpopular (Rogers, 2012). It is critical to have advocacy skills and credibility (Joyce et al., 2014). Nurses have individual as well as group identities and ideals. The purpose of this research was to see how an interactive digital-based training program affected primary healthcare rural nurses' understanding, self-efficacy, and environmental activism in the context of climate change.

DETAILED DESCRIPTION:
The threat of climate change to human health and survival is significant (Watts et al. 2019). The planet has warmed by over 1.2°C since preindustrial times; causing severe and rapidly deteriorating health affects worldwide (Butterfield et al., 2021). Despite overwhelming evidence, however, the global response to climate change has been hindered by political intransigence and bureaucracy. Health professionals are increasingly looked to for leadership and their continued commitment is addressing critical gaps in climate science, policy, and advocacy (Watts et al. 2020).

The environment plays a vital role in determining human health (Anderko et al., 2014; Nichols et al., 2009). A direct link exists between climate change and air pollution, which takes the lives of over 7 million people each year (World Health Organization, 2018). Nurses worldwide have expressed deep concerns about sustainability (Dunphy, 2014). Some nurses are now becoming environmental activism. Fielding et al. (2008, p.219) define "environmental activism" as "purposeful and effortful engagement in behaviors aimed at preserving or improving the quality of the environment and increasing public awareness of environmental issues and may include protesting, rallying, petitioning, educating the public, lobbying government and corporations, participating in direct actions such as blockades or participating in voluntary conservation or revegetation work." Perceived self-efficacy, the degree to which people believe they are capable of performing specific tasks to achieve certain goals, is a central concept in Bandura's Social Cognitive Theory (Bandura, 2011; Schunk, 2013). It impacts individuals through four main processes: selection, motivational, affective, and cognitive dimensions. Grothmann and Patt (2005) propose two cognitive appraisal processes that people would undertake to protect themselves and adapt to climate change impacts. These are "risk appraisal-the perceived probability of being exposed to risk and its perceived severity; and adaptation appraisal-the ability to avert being harmed by the threat, along with the costs of taking such action, which results in an awareness of perceived adaptive capacity" (Grothmann & Patt, 2005). Regardless of whether an individual perceives some threats to be low or high, they will engage in appraising their efficacy (Witte, 1992; Witte, 1998). However, those who perceive or believe the threats or hazards to be high are more likely to take protective action to avert harm.

Self-efficacy is an individual's belief in their capacity to execute behaviors necessary to reduce or prevent damage (Witte, 1998; Bandura, 1997). Perceived self-efficacy reflects confidence in the ability to exert control over one's own behavior and social environment, making it crucial in understanding human behavior (Hanson-Easey, 2013). While self-efficacy is increasingly being used to understand human responses to climate change, its use has been mainly restricted to studies on mitigation rather than adaptation. Self-efficacy potentially determines whether an individual will adapt or not, and it also determines the nature of transformation and how an individual will adapt to climate change.

The impact of climate change on humans has become one of the most prominent issues on the international agenda in recent decades. Climate change implications vary within and between locations due to multiple factors, including physical features, coping capacities, and sensitivities (Folke, 2006; Smit et al., 2006). Climate change mitigation and adaptation have emerged in the climate change discourse. While the former aims to avoid the unmanageable, the latter aims to manage the unavoidable (Huang et al., 2011). Although mitigation dominated international climate policy discussions in the 1990s and early 2000s, lately, growing attention (in both theory and practice) is being given to adaptation. Adaptation to climate change has become a prominent topic of current policy development and debates (Adger, 2006; Adger et al., 2009). According to Smit and Pilifosova (2003), "adaptation is important in climate change response in two ways: the assessment of impacts and vulnerabilities and the development and evaluation of response options." Given the pace at which the climate changes and the potential adverse impacts, adaptation "is no longer tomorrow's choice, but today's imperative" (Huang et al., 2011). In developing countries, where high dependency on climate-sensitive natural resources and the elevated impact of climate change persist, adaptation has been one of the focal points of current development discussions (Barros, 2014).

Information and communication technologies (ICT) have evolved to be typical in modern life. The use of modern communication technologies in healthcare is expanding access to healthcare services and expanding resource availability, especially among underprivileged groups. Digital technologies are said to improve healthcare providers communication, encourage laypeople to participate in preventative health activities, and improve adherence to treatment regimens. It is gaining popularity as proof of its usefulness in increasing awareness about climate change (Lupton, 2013). Furthermore, digital-based education may provide individualised and personalised teaching, feedback, and goal setting, improving client-centered care and communication and training individuals with little understanding of climate change to improve their knowledge and attitude (SRI, 2018).

The nursing profession was an early participant in the climate change discussion and is well-positioned to increase its involvement. Nurses have three valuable assets. First, they account for over 60% of all health professionals worldwide, operating in a variety of clinical and public health settings (WHO, 2020). Their collective power to alter the course of climate action is unrivalled. Nurses have an important role and can be more effective communicators of the moral tale of climate change. They have a history of defending human dignity, and the public feels at ease with nurses discussing what is right and wrong. Nursing should enhance its commitment to climate-friendly indigenous practices and ancestral knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. being 20 years or older,
2. owning a smartphone,
3. being willing to participate in the study.
4. Both male and female nurses.

Exclusion Criteria:

1 - Not able to use Smartphones.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Climate change/global warming knowledge questionnaire | through study completion, an average of 1 year
  It is a measure of knowledge regarding global warming and climate change, and related consequences, developed by Salem et al. (2022). The questionnaire is valid and reliable, with Cronbach's alpha coefficient of 0.879. It comprises 15 questions that are answered by either yes= 1 or no=0 or I don't know=0. The knowledge percent score was grouped as knowledgeable ≥70%, not knowledgeable <70%.

SECONDARY OUTCOMES:
Environmental self-efficacy scale (ESE) | through study completion, an average of 1 year
  Environmental self-efficacy scale (ESE) developed by Bryton & Alexander (2019). It is used to measure environmental self-efficacy. It consists of 20 items rated on a 11-point Likert scale, with 0 denotes cannot do at all, and 10 denotes highly certain can do, with higher scores indicating higher environmental self-efficacy. It includes items related to specific types of ESE, and barriers of ESE.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Hashem El-Monshed, Al Mansurah, Dakhlyia, Egypt

IPD SHARING:
Plan to Share IPD: No